CLINICAL TRIAL: NCT03346369
Title: Lanthanum Carbonate (Fosrenol®) to Reduce Oxalate Excretion in Patients With Secondary Hyperoxaluria and Nephrolithiasis: a Short-term, Prospective, Open-label, Efficacy and Safety Clinical Trial
Brief Title: Lanthanum Carbonate (Fosrenol®) to Reduce Oxalate Excretion in Patients With Secondary Hyperoxaluria and Nephrolithiasis
Acronym: LaCa
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: oxalate01
Record Dates: First submitted 2017-03-28; First posted 2017-11-17 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Secondary Hyperoxaluria; Nephrolithiasis
Keywords: Nephrolithiasis; Urolithiasis; Secondary Hyperoxaluria; Hyperoxaluria; Lanthanum Carbonate; Phosphate Binder
MeSH Terms: conditions — Nephrolithiasis; Urolithiasis; Hyperoxaluria | interventions — lanthanum carbonate

STUDY DESIGN:
Intervention Model Description: This study investigates the efficacy and the safety of Lanthanum Carbonate for the reduction of urinary oxalate excretion in patients with secondary hyperoxaluria and nephrolithiasis. Patients will be treated during 2 consecutive 14-day treatment periods with a low and a high dose of Lanthanum Carbonate respectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental single arm (Experimental): Treatment with Lanthanum Carbonate 3 x 250 mg/day with meals during a first 14-day treatment period. Subsequently, treatment with Lanthanum Carbonate 3 x 500 mg/day with meals during a second 14-day treatment period.
  Interventions: Drug: Lanthanum Carbonate

INTERVENTIONS:
Drug: Lanthanum Carbonate — Treatment with Lanthanum Carbonate 3 x 250 mg/day with meals during a first 14-day treatment period. Subsequently, treatment with Lanthanum Carbonate 3 x 500 mg/day with meals during a second 14-day treatment period

SUMMARY:
This study investigates the efficacy and the safety of Lanthanum Carbonate for the reduction of urinary oxalate excretion in patients with secondary hyperoxaluria and nephrolithiasis.

DETAILED DESCRIPTION:
Nephrolithiasis/urolithiasis is a prevalent (overall lifetime risk up to 13% in Western countries) and highly recurrent disease. Secondary hyperoxaluria is a key risk factor for the development of calcium oxalate stones, the most frequent stone type. Currently used therapeutic options in secondary hyperoxaluria have limited efficacy. Recent findings in vitro and in a rat model, provided evidence that Lanthanum Carbonate is an effective oxalate binder. The objective of this study is to investigate whether treatment with Lanthanum Carbonate reduces urinary oxalate excretion in human subjects with secondary hyperoxaluria and nephrolithiasis. By treating the patients with two different doses of Lanthanum Carbonate during two 14-day treatment periods, a dose-response will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* able to give written informed consenct
* hyperoxaluria (defined as urinary oxalate > 45 mg/24 hours), demonstrated on 24-hour urine collection within 18 months prior to baseline visit
* history of nephrolithiasis eGFR > 60 mL/min/1.73m² (CKD-EPI formula)

Exclusion Criteria:

* primary hyperoxaluria, diagnosed by genetic testing
* known allergy to Lanthanum Carbonate
* hypophosphatemia (defined as serum phosphorus < 0.81 mmol/L)
* severe known liver insufficiency of biliary obstruction
* rectocolitis ulcerohaemorraghica, Crohn's disease, bowel obstruction, stomach/duodenal ulceration
* glucose/galactose malabsorption
* severe diarrhea or other gastrointestinal disorder, which might interfere with the ability to absorb oral medication
* pregnancy or breast-feeding
* female participant of childbearing potential unwilling to take efficient contraceptive measures for the duration of the study
* female participant without negative serum or urine pregnancy test
* psychological illness or condition, interfering with the patient's compliance or ability to understand the requirements of the study
* currently participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2017-08-18 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The mean reduction in urinary oxalate excretion in patients treated with a daily Lanthanum Carbonate dose of 750 mg | After the first 14-day treatment period
  Mean reduction in urinary oxalate excretion after the first 14-day treatment period during which patients will be treated with 250 mg Lanthanum Carbonate 3x/day with meals, expressed in mg oxalate/g creatinine.

SECONDARY OUTCOMES:
The incremental reduction in mean urinary oxalate excretion after doubling the dose of Lanthanum Carbonate from 750 mg tot 1500 mg daily | After the second 14-day treatment period
  Incremental reduction of mean urinary oxalate excretion after the second 14-day treatment period during which the patients will be treated with 500 mg Lanthanum Carbonate 3x/day with meals, expressed in mg oxalate/g creatinine
The proportion of patients developing severe hypophosphatemia | After the first and second 14-day treatment period
  Severe hypophosphatemia is defined as serum phosphorus < 0.64 mmol/L
The evolution of phosphaturia, evaluated by 24-hour urinary phosphorus excretion | After the first and second 14-day treatment period
  24-hour urinary phosphorus excretion will be expressed in mmol/24 hours
The evolution of phosphaturia, evaluated by urinary phosphorus to creatinine ratio | After the first and second 14-day treatment period
  Urinary phosphorus to creatinine ratio will be expressed in mmol phosphorus/g creatinine
The evolution of phosphaturia, evaluated by fractional excretion of phosphorus | After the first and second 14-day treatment period
  Fractional excretion of phosphorus will be expressed in %, defined as (urinary phosphorus (mmol/L) x serum creatinine (mg/dL) / (serum phosphorus (mmol/L) x urine creatinine (mg/dL))
The proportion of patients developing hypophosphaturia | After the first and second 14-day treatment period
  Hypophosphaturia is defined as urinary phosphorus < 12.9 mmol/24 hours
The evolution of calciuria, evaluated by 24-hour urinary calcium excretion | After the first and second 14-day treatment period
  24-hour urinary calcium excretion will be expressed in mmol/24 hours
The evolution of calciuria, evaluated by urinary calcium to creatinine ratio | After the first and second 14-day treatment period
  Urinary calcium to creatinine ratio will be expressed in mmol calcium/g creatinine
The evolution of calciuria, evaluated by fractional excretion of calcium | After the first and second 14-day treatment period
  Fractional excretion of calcium will be expressed in %, defined as (urinary calcium (mmol/L) x serum creatinine (mg/dL)) / (serum calcium (mmol/L) x urine creatinine (mg/dL))
The evolution of serum Lanthanum levels | After the first and second 14-day treatment period
  Serum Lanthanum levels will be expressed in mcg/L
Adverse events | After the first and second 14-day treatment period
  The number and the proportion of patients experiencing adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Christian Tielemans, MD, PhD, Principal Investigator — Department of Nephrology, University Hospital Brussels
Locations (1):
- University Hospital Brussels, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No